CLINICAL TRIAL: NCT02336269
Title: Protocol For The Evaluation of Primex's PGX Assay
Brief Title: Evaluation of Primex's PGX Assay to Assess the Clinical Utility of Pharmacogenomics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Primex Clinical Laboratories, Inc. (Industry)
Collaborators: Research & Development Institute, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RDI-PGX-80801.01
Record Dates: First submitted 2015-01-05; First posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Patients on Medications Metabolized Via CYP450
Keywords: Pharmacogenomics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swab
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Primex's PGX assay is an in vitro, semi automated assay, intended for the determination of certain genes involved in drug metabolism utilizing buccal swabs. Detection of certain genotypes is used as an aid in the selection of appropriate medications based on the individuals' specific genotype and should be used in conjunction with other clinical information. The results from this tests constitutes one parameter in a multicriterion medication selection process, encompassing both clinical and laboratory-based assessments.

DETAILED DESCRIPTION:
The way a person responds to a drug (this includes both positive and negative reactions) is a complex trait that is influenced by many different genes. Without knowing all of the genes involved in drug response, scientists have found it difficult to develop genetic tests that could predict a person's response to a particular drug. Once scientists discovered that people's genes show small variations (or changes) in their nucleotide (DNA base) content, all of that changed-genetic testing for predicting drug response is now possible. Pharmacogenomics is a science that examines the inherited variations in genes that dictate drug response and explores the ways these variations can be used to predict whether a patient will have a good response to a drug, a bad response to a drug, or no response at all.

The Gene super family of Cytochrome P450 is primarily responsible for clearance of the different drugs and variations in different genes affect the metabolism of different classes of drugs. In our test we have concentrated on the genes and specific variations of those genes which have been studied best and already have existing and convincing data by peer reviewed journals.

Since one of the major classes of drugs that are affected by the Cytochrome P450 pathway are anti-coagulants, we have also added certain genes that are involved in coagulation variations of which might have additive affects on the coagulation status of the patient. Having this information can aid the physician in making better decisions when prescribing or dosing anti-coagulants.

Description of the Primex PGX Assay:

DNA is isolated from subject buccal swabs and is subjected to PCR and Real Time PCR for determination of the genetic variations detailed above. After the variations are determined, known effects of the variations (i.e. reduced activity or hyperactivity) are reported to a pharmacist and these effects in combination with the subjects medication list are used to further establish clinical significance or utility. The physician then can make a decision to change the medication as recommended. If the physician makes any changes to the subject's medication regimen, then in 3 months he/she will assess the changes and reports the findings; hence establishment of the clinical utility of our test.

Analytical Performance Objectives:

Assess the reproducibility of Primex's PGX assay with samples run in replicates of 3, twice a day, for a minimum 5 days.

Clinical Performance Evaluation Objectives:

Assess the clinical performance characteristics of Primex's PGX assay for the genotypes determined in the different genes of the CYP450 gene super family and genes related to coagulation by Life Technology's QuantSudio 12kFlex open array real time PCR system. There are no predicate devices therefore the clinical utility will be assessed by predicted phenotype and the number of effective changes made by the physicians to the subject's drug regimen.

Acceptance criteria for comparison of the Primex's PGX assay results to clinical changes made to the subject's drug regimen:

The clinical sensitivity and specificity of the Primex's PGX assay results to clinical changes made are a minimum of 65% and 90%, respectively. Results of the prior drug regimen changes before Primex's PGX testing will be provided and may be used for comparative analysis.

Investigator Feedback:

At the conclusion of the clinical study, the investigator will assess the clinical performance characteristics evaluated and acceptability of the Primex's PGX assay in a written report/letter to the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Buccal swab sample prospectively collected under Informed Consent
* Remnant Buccal swab sample meeting the FDA requirements for use of leftover specimen
* Samples from at least one of the following groups:
* specimens from subjects who are on multiple medications of which at least 2 are affected by the pathways tested and the physician made changed to their drug regimen based on the assay interpretations
* subjects who are on multiple medications of which at least 2 are affected by the pathways tested and the physician made no changes based on the assay interpretations
* Subjects with Chronic disease
* Subjects with different ethnic backgrounds
* Subjects from different geographical areas
* Apparently healthy subjects
* Clinical information required per CRF is available

Exclusion Criteria:

- Samples that do not meet all inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A minimum of 10,000 buccal swab samples will be identified for inclusion in the study as follows:
  * A minimum of 8700 specimens from subjects who are on multiple medications of which at least 2 are affected by the pathways tested and the physician made changed to their drug regimen based on the assay interpretations
  * A minimum of 5200 specimens from subjects who are on multiple medications of which at least 2 are affected by the pathways tested and the physician made no changes based on the assay interpretations
  * A minimum of 1100 apparently healthy subjects.
  Study subjects may be enrolled prospectively, from collection sites.
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Clinical Utility of Primex's PGX assay as measured by medication change/no-change by the physician based on Primex's PGX assay results as an aid in the prediction of drug response | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Research and Development Institute, Van Nuys, California, United States